CLINICAL TRIAL: NCT01135706
Title: Fractal Analysis of the Pulmonary Arterial Tree in Pulmonary Hypertension.
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Karen Wood, M.D., Ohio State University
Other Study IDs: 2010H0097
Record Dates: First submitted 2010-05-20; First posted 2010-06-03 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Fractal dimension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pulmonary Hypertension: Patients having a right heart catheterization and CT pulmonary angiogram with a diagnosis of Pulmonary Hypertension
  Interventions: Other: No Intervention
- Non Pulmonary Hypertension: Patients having a right heart catheterization and CT pulmonary angiogram without a diagnosis of Pulmonary Hypertension.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This study does not include an intervention but is observational in nature.

SUMMARY:
The investigators propose to confirm that normotensive and hypertensive pulmonary arteries are fractal, as well as define if the FD correlates to disease severity when compared to available data such as six-minute walk and right heart catheterization measurements.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is an insidious disorder that can occur in isolation or as a result of various other pulmonary and systemic conditions. If left untreated PH may progress to right heart failure and death. Numerous tests are suggestive but not diagnostic of PH including cardiac echo, pulmonary function testing and chest x-ray. Definitive diagnosis requires right heart catheterization that is invasive, costly and time consuming. The fractal dimension (FD) is an index of the space-filling properties of an object so that the closer the dimension is to the topological dimension in which the object is embedded, the greater the space filling properties. No investigations have been performed to analyze the fractal dimension of pulmonary arteries in patients with PH. We propose to confirm that normotensive and hypertensive pulmonary arteries are fractal, as well as define if the FD correlates to disease severity when compared to available data such as six-minute walk and right heart catheterization measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a right heart catheterization and CT pulmonary angiogram

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a right heart catheterization and CT pulmonary angiogram
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
FD of the pulmonary artery in patients with PH will be lower when compared to patients without PH. | 24 Months

SECONDARY OUTCOMES:
FD will correlate with the degree of PH as quantified by the MPAP obtained during RHC. | 24 Months
FD will correlate with the functional capacity of the PH patients as quantified by distance during six-minute walk and NYHA functional class. | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Wood, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States